CLINICAL TRIAL: NCT02211885
Title: A Phase I Single Oral Dose (100 mg) Trial to Characterize the Excretion Balance of 14c-radiolabeled BIRB 796 BS and to Determine Its Metabolites in Normal Male Subjects
Brief Title: Excretion Balance of 14c-radiolabeled BIRB 796 BS in Normal Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1175.6
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: 14C-BIRB 796 BS — 14C-radiolabeled BIRB 796 BS

SUMMARY:
Study to characterize the pharmacokinetics of 14C-radiolabeled BIRB 796 BS and its metabolites including excretion and mass balance of parent compound and radioactivity; to isolate, identify and quantify major radiolabeled metabolites of BIRB 796 in plasma, urine and feces

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening. Health is confirmed by medical history, physical examination, laboratory testing and 12-lead electrocardiogram (ECG)
* Signed written informed consent in accordance with Good Clinical Practice
* Age ≥ 18 and ≤ 45 years
* Subjects within 10% of the normal height: weight range defined by the Metropolitan Life Insurance Company Tables

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and ECG) deviating from normal and of clinical relevance
* History of clinically significant disease including metabolic, endocrinologic, immunological, hepatic, renal, gastrointestinal, respiratory, cardiovascular, psychiatric or neurological
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Subjects with a history of drug abuse or alcoholism
* Chronic or relevant acute (within 1 month of screening) infections
* Subjects who have taken prescription within one month or over-the-counter drugs within two weeks of the start of the trial
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during trial)
* Inability to refrain from smoking on trial days
* Blood donation > 400 mL (within 1 month prior to administration or during the trial)
* Any laboratory value outside 10% of the reference range of clinical relevance (but not exclusive to) total white cell count ≥ 10 x 10**9/L, any hemoglobin < 12 mg/dl or >15 mg/dl. Protein on urine dipstick
* Positive urine drug screen, positive HIV or Hepatitis C antibodies
* History of any familial bleeding disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2002-10; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Cumulative amount of 14C-BIRB 796 BS radioactivity excreted in feces (percent of dose) | up to 5 days
Cumulative amount of 14C-BIRB 796 BS radioactivity excreted in urine (percent of dose) | up to 5 days
Maximum observed Concentration (Cmax) of 14C-BIRB 796BS in plasma | up to 96 hours after drug administration
Area under the Concentration versus time curve from time 0 to infinity (AUC0-∞) of 14C-BIRB 796BS in plasma | up to 96 hours after drug administration
Time To The Maximum Concentration (tmax) of 14C-BIRB 796BS in plasma | up to 96 hours after drug administration
Elimination Half-Life (t1/2) of 14C-BIRB 796BS in plasma | up to 96 hours after drug administration
Erythrocyte-plasma partition ratio of 14C-radioactivity | up to 5 days
Cmax of 14C-BIRB 796BS in blood | up to 96 hours after drug administration
AUC0-∞ of 14C-BIRB 796BS in blood | up to 96 hours after drug administration
tmax of 14C-BIRB 796BS in blood | up to 96 hours after drug administration
t1/2 of 14C-BIRB 796BS in blood | up to 96 hours after drug administration
Cmax of BIRB 796BS in plasma | up to 96 hours after drug administration
AUC0-∞ of BIRB 796BS in plasma | up to 96 hours after drug administration
tmax of BIRB 796BS in plasma | up to 96 hours after drug administration
t1/2 of BIRB 796BS in plasma | up to 96 hours after drug administration
Quantification of radiolabeled metabolites in urine (percent of dose) | up to 5 days
Quantification of radiolabeled metabolites in feces (percent of dose) | up to 5 days
Quantification of radiolabeled metabolites in plasma (percent of dose) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
Excretion of 14C-radioactivity in saliva (percent of dose) | up to 24 hours after drug administration
Excretion of 14C-radioactivity in expired air (percent of dose) | up to 48 hours after drug administration